CLINICAL TRIAL: NCT01264068
Title: The Influence of Chinese Medicine on Metabolomics in Menopausal or Postpartum Women
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei City Hospital (Other Government)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Jung-Lien Lai/Taipei City Hospital, Taipei City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TCHIRB-970208-E
Record Dates: First submitted 2010-12-20; First posted 2010-12-21 (Estimated); Last update posted 2010-12-21 (Estimated); Status verified 2008-03

CONDITIONS: Menopausal Women
Keywords: Suan-Tsao-Jen-Tang ,Jia-Wey-Shiau-Yau-San,metabolomics,menopause

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Insomnia control (No Intervention)
- Suan Tsao Jen Tang (Experimental)
  Interventions: Drug: Finished Herbal Product such as Suan Tsao Jen Tang, Jia-Wey Shiau-Yau San
- Jia-Wey Shiau-Yau San (Experimental)
  Interventions: Drug: Finished Herbal Product such as Suan Tsao Jen Tang, Jia-Wey Shiau-Yau San

INTERVENTIONS:
Drug: Finished Herbal Product such as Suan Tsao Jen Tang, Jia-Wey Shiau-Yau San — Take medicine every day 3 times, each time 4 grams.
  Arms: Jia-Wey Shiau-Yau San; Suan Tsao Jen Tang

SUMMARY:
Traditional Chinese herbal medicine, no matter mono-therapy or poly-pharmacy, is composed of complicated chemical constituents. Many confounding factors influence activity of Chinese herbs, including the origin of the herbs, safety of the products and consistency between batches. Study of the effectiveness and mechanism of Chinese herbs in vivo is much more challengeable due to unresolved problems of product quality control, screen of effective principles, monitor of the marker constituents and the targets for site of action. In this project, we will introduce the concept of metabolomics to detect total metabolites spectra as the biomarkers of Chinese herbs intervention. Correlation will be analyzed between changes in total metabolites and clinical improvements when menopausal women receive Suan Tsao Jen Tang or Jia Wey Shiau Yau San, and postpartum women receive生化湯.

ELIGIBILITY:
Inclusion Criteria:

* Insomnia according to PSQI>6
* Informed consent
* Female
* Age 40-65 years

Exclusion Criteria:

* In 3 months before participating in and studying, happen great accident or heavy night shift or have time difference problems (such as the long-range flight) .
* Spiritual disease (melancholia,etc.) ,obstructive sleep apnea, heart disease history (the acute heart attack, cardiac arrhythmia) , hypertension , diabetes mellitus, cancer.
* Take melatonin or melatonin agonist, such medicines as acetylcholine, glutamate, serotonin, norepinephrine, GABA, histamine, adenosine, prostaglandins,etc..

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-04 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Total metabolites detection using LC/MS/MS | one month

SECONDARY OUTCOMES:
1.Menopause rating scale (MRS) 2.Pittsburgh sleep quality index (PSQI) | one month

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Hui Chen, PHD, Study Chair — Associate Professor, School of Pharmacy,National Taiwan University
Locations (1):
- Taipei City Hospital, Taipei, Taiwan, Taiwan